CLINICAL TRIAL: NCT01897506
Title: Assessing Risk of Food Insecurity Within Households of Children With Food Allergy
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 201920
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Food Allergy; Asthma; Allergic Rhinitis; Atopic Dermatitis; Eosinophilic Esophagitis
Keywords: Food insecurity; Health literacy; Quality of life
MeSH Terms: conditions — Food Hypersensitivity; Asthma; Rhinitis, Allergic; Dermatitis, Atopic; Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our central hypothesis is that dietary limitations introduced by food allergy will contribute to increased food insecurity in households with food allergic children when compared to food insecure households without food allergic children.

DETAILED DESCRIPTION:
Specific Aim 1 To describe food insecurity in families of the pediatric allergy population, specifically comparing the prevalence of food insecurity rates between households of food allergic patients and households of allergic patients without food allergy.

Specific Aim 2 To examine health literacy in parents of patients in the pediatric allergy population, comparing food insecure patients with and without food allergy to food secure patients with food allergy.

Specific Aim 3 To examine quality of life in food allergic patients' households using the food allergy impact scale, comparing food allergic patients' households with food insecurity to food allergic patients' households without food insecurity.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose child has an allergy appointment with the Allergy and Immunology Department at Arkansas Children's Hospital between 1-17 years of age with allergic disease

Exclusion Criteria:

* Parents whose child has an allergy appointment with the Allergy and Immunology Department at Arkansas Children's Hospital less than 1 years of age or 18 years of age and older will not be eligible to participate in this study. Children with immunodeficiency disease will be excluded.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Families with children who have allergy appointments at Arkansas Children's Hospital between 1-17 years of age. We will recruit 325 families with patients in the food allergy group and 325 families with patients in the without food allergy group.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Presence of food insecurity within an atopic population | 1.25 years
  The primary outcome variable of interest is the presence of food insecurity (patients with Low Food Security or Very Low Food Security). A chi-square test of independence will be used to test the association between food insecurity and food allergy.

SECONDARY OUTCOMES:
Health Literacy Rate | 1.25 years
  A logistic regression analysis will be done to test the effect of food allergy and food insecurity on the health illiteracy rates after adjusting for confounding variables such as demographics. Appropriate contrasts for the interaction effect between food allergy and food insecurity will also be used to compare health literacy rates.

OTHER OUTCOMES:
Quality of life of families with food allergic members | 1.25 years
  The average quality of life score taken across all six items in the quality of life questionnaire will be the outcome variable of interest. The mean average quality of life score between the food secure households with food allergy and the food insecure households with food allergy will be compared between the two groups using an ANCOVA method.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie M Jones, MD, Principal Investigator — University of Arkansas for Medical Sciences / Arkansas Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States